CLINICAL TRIAL: NCT00427726
Title: Follow-Up Study of Breast Cancer and Multiple Myeloma Subjects Previously Enrolled in Retroviral Gene Transfer Studies
Brief Title: Follow-up of Breast Cancer and Multiple Myeloma Patients Previously Enrolled in NIH Gene Therapy Studies
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030124; 03-C-0124; NCT01444937 (obsolete NCT alias)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-05-20

CONDITIONS: Gene Transfer
Keywords: Gene Transfer; Hematopoietic Stem Cells; Follow-Up

SUMMARY:
This study will provide follow-up evaluations of breast cancer or multiple myeloma patients who received gene therapy (gene transfer) as part of their participation in an NIH protocol. Gene therapy is a new technology, which may involve a permanent change in the patient s genetic code. Therefore, although the risk of long-term harmful effects of this therapy is very small, the Food and Drug Administration requires prolonged monitoring of patients health status.

Patients previously enrolled in NIH protocols 96-C-0007, 93-C-0208, 92-C-0161, or 92-H-0057 will be followed under the current protocol. No further gene therapy will be provided in this study.

Patients health status will be evaluated for an indefinite period of time, or as long as they are willing to be monitored. They will provide a blood sample once a year and will be interviewed about their health status twice a year for the first 5 years after gene therapy and once a year thereafter. These procedures are done to look for the development of any diseases such as cancer, neurological disorders, autoimmune or blood disorders that may be related to side effects of the gene transfer.

DETAILED DESCRIPTION:
This Protocol aims to provide long-term follow-up of breast cancer and multiple myeloma subjects previously receiving autologous primitive marrow and blood hematopoietic cells exposed to gene transfer retroviral vectors on the following protocols: MB 294 (92-C-0161; T-92-0018), MB 310 (93-C-0208; T-92-0192), MB 361 (96-C-0007; T-95-0096) or (92-H-0057; T-92-0139) at the National Cancer Institute and the National Heart, Lung, and Blood Institute. Subjects will undergo an annual health history and annual complete blood counts will be performed. Blood samples will also be collected annually (either locally or off-site by the subjects' personal physicians) for testing for presence of the gene transfer vector and vector integration sites.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who received gene transfer products on the following protocols: MB 361, 96-C-0007, T-95-0096; MB 294, 92-C-0161, T-92-0018; MB 310, 93-C 0208, T-92-0192; or 92-H-0057, T-92-0139.

EXCLUSION CRITERIA:

Patients unwilling to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-03-06; Study Completion 2014-05-20

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dunbar CE, Cottler-Fox M, O'Shaughnessy JA, Doren S, Carter C, Berenson R, Brown S, Moen RC, Greenblatt J, Stewart FM, et al. Retrovirally marked CD34-enriched peripheral blood and bone marrow cells contribute to long-term engraftment after autologous transplantation. Blood. 1995 Jun 1;85(11):3048-57. PMID 7538814
- [Background] Cowan KH, Moscow JA, Huang H, Zujewski JA, O'Shaughnessy J, Sorrentino B, Hines K, Carter C, Schneider E, Cusack G, Noone M, Dunbar C, Steinberg S, Wilson W, Goldspiel B, Read EJ, Leitman SF, McDonagh K, Chow C, Abati A, Chiang Y, Chang YN, Gottesman MM, Pastan I, Nienhuis A. Paclitaxel chemotherapy after autologous stem-cell transplantation and engraftment of hematopoietic cells transduced with a retrovirus containing the multidrug resistance complementary DNA (MDR1) in metastatic breast cancer patients. Clin Cancer Res. 1999 Jul;5(7):1619-28. PMID 10430060
- [Background] Emmons RV, Doren S, Zujewski J, Cottler-Fox M, Carter CS, Hines K, O'Shaughnessy JA, Leitman SF, Greenblatt JJ, Cowan K, Dunbar CE. Retroviral gene transduction of adult peripheral blood or marrow-derived CD34+ cells for six hours without growth factors or on autologous stroma does not improve marking efficiency assessed in vivo. Blood. 1997 Jun 1;89(11):4040-6. PMID 9166843